CLINICAL TRIAL: NCT05160688
Title: Changes in Cognition and Psychiatric Disorder Symptoms During Cannabis Abstinence Using a Novel Discordant Twin Design
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Colorado, Boulder (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21-4899
Record Dates: First submitted 2021-11-19; First posted 2021-12-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Cannabis
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingency management (Experimental): Contingency management (CM) is an incentive-based intervention providing patients with tangible rewards as reinforcement for positive behaviors like abstinence from drug use. Incentives are provided with each urine sample that is drug-free and are increased with each subsequent drug-free urine sample. Participants in the CM condition will receive increasing payments for abstinence: $30 on day 3, $45 on day 5, $60 on day 7, $75 on day 14, $90 on day 21, $105 on day 28, and $120 on day 42. Participants in both conditions also receive increasing payment for visit attendance: $10 on day 1, $15 on day 3, $20 on day 5, $25 on day 7, $30 on day 14, $35 on day 21, $45 on day 28, and $55 on day 42. At the end of the baseline visit, participants in the CM condition will sign a behavioral contract with study staff that clearly outlines expectations as well as the payment schedule.
  Interventions: Behavioral: Contingency management
- No intervention (No Intervention): Participants in this condition will be monitored and will not receive any compensation for cannabis abstinence.

INTERVENTIONS:
Behavioral: Contingency management — Participants will be paid to abstain from cannabis use.
  Arms: Contingency management

SUMMARY:
This study will test whether 42 days of cannabis abstinence, compared to continued cannabis use, is associated with improvements in cognition and psychiatric disorder symptoms. Identical twins, who are concordant on cannabis use, will be experimentally-manipulated to be discordant for 42 days. Each twin, within a twin pair, will be randomly assigned to either the contingency management condition, incentive-based protocol to promote cannabis abstinence, or control condition, no changes in cannabis use requested.

DETAILED DESCRIPTION:
The proposed project is a randomized controlled trial to compare cognition and psychiatric disorder symptoms between monozygotic (MZ) twin pairs, who are concordant on frequency of cannabis use. Each twin, within the twin pair, will be randomly assigned to either contingency management (CM), monetary incentives provided to reinforce cannabis abstinence, or control, no changes in cannabis use required or reinforced. Participants in the CM condition will receive an increasing schedule of payments at each visit reinforcing continued cannabis abstinence. All participants will receive increases in the payment schedule for attendance of each subsequent assessment. Participants will be assessed on measures of cognition including attention, memory, and processing speed as well as anxiety, depression, and ADHD symptoms. In addition, at each visit participants will complete a qualitative and quantitative drug test. The qualitative drug test will be used to determine if new cannabis use has occurred since the last visit, and will determine if the participant receives payment for abstinence. The investigators will also use previously collected genotype for each participant.

The first aim of this study is to characterize cognitive recovery, across all potential cognitive domains, using an experimental manipulation to achieve discordance between MZ twins on cannabis use. The hypothesis for the first aim is that the abstinent group will have greater improvements in memory and processing speed compared to controls. However, there will not be any group differences between the abstinent group and the control group on attention, language, and executive function performance. The second aim of the proposed project is to characterize psychiatric disorder symptoms by comparing psychiatric disorder symptom changes among the cannabis abstaining twin to their cannabis using co-twin across 42 days. The abstinent group will endorse more psychiatric symptoms during the withdrawal period (up to 14 days) but will endorse fewer psychiatric symptoms at day 28 and 42 compared to the control group. The third aim (exploratory) of the proposed project is to examine how genetic risk for psychiatric disorders interacts with environment (i.e., cannabis abstinence versus continued use) to influence cognitive functioning. The hypothesis for aim 3 is that anxiety, depression, and ADHD polygenic scores will be more strongly associated with cognitive outcomes in the control group compared to the abstinent group.

ELIGIBILITY:
Inclusion Criteria:

1. Monozygotic (MZ) twin pair, in which both twins are willing to participate
2. MZ twin pair must be concordant in their frequency of cannabis use (+/- 2 days)
3. Cannabis use at least 1x per week on most weeks
4. Cannabis use in the past 7 days at the baseline visit
5. Positive qualitative urine toxicology at baseline for THC
6. Located within the state of Colorado

Exclusion Criteria:

1) Discordance in the twin pairs on a significant, adverse experience, like traumatic brain injury.

Ages: 31 Years to 47 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in attention performance | Change from baseline to day 42
  Flanker Inhibitory Control and Attention Test on NIH Toolbox: Composite score of accuracy and reaction time
Change in episodic memory | Change from baseline to day 42
  Picture Sequence Memory Test on NIH Toolbox: Cumulative number of correct adjacent pairs
Change in working memory | Change from baseline to day 42
  List Sorting Working Memory Test on NIH Toolbox: Total items correct across all trials
Change in receptive vocabulary | Change from baseline to day 42
  Picture Vocabulary Test on NIH Toolbox: Computer adaptive testing
Change in reading decoding | Change from baseline to day 42
  Oral Reading Recognition Test: Number of letters and words read correctly
Change in immediate memory/verbal learning | Change from baseline to day 4
  Auditory Verbal Learning Test on NIH Toolbox: Total number of words recalled
Change in pattern comparison processing speed | Change from baseline to day 42
  Pattern Comparison Processing Speed Test: Total number of correct responses
Change in oral symbol digit test processing speed | Change from baseline to day 42
  Oral Symbol Digit Test on NIH Toolbox: Total number of correctly identified symbols
Change in attention and executive function | Change from baseline to day 42
  Dimensional Change Card Sort Test on NIH Toolbox: Composite score of accuracy and correct answers

SECONDARY OUTCOMES:
Change in anxiety symptoms | Change from baseline to day 42
  Beck Anxiety Inventory: Total score. Scores range from 0-63 and higher scores indicate higher levels of anxiety.
Change in depressive symptoms | Change from baseline to day 42
  Beck Depression Inventory: Total score. Scores range from 0-63 and higher scores indicate greater levels of depression.
Change in attention deficit/hyperactivity disorder symptoms | Change from baseline to day 42
  Adult Self-Report Scale: Total score. Scores range from 0-72 and higher scores indicate greater level of symptoms of attention deficit/hyperactivity disorder.

CONTACTS AND LOCATIONS:
Overall Officials: J. Megan Ross, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- Jessica M Ross, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
In accordance with NIH data sharing policies, data produced from this project will be made available to ensure timely translation of research results to improve human health. The investigators believe there is a possibility of deductive disclosure of subjects with unusual characteristics, even though all identifiers would be removed prior to release for sharing. Thus, the investigators will make the data and associated documentation available to users only under a specific data-sharing agreement that requires: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.